CLINICAL TRIAL: NCT05263999
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Multicenter Study of Itolizumab in Combination With Corticosteroids for the Initial Treatment of Acute Graft Versus Host Disease
Brief Title: A Study of Itolizumab in Combination With Corticosteroids for the First-Line Treatment of Acute Graft Versus Host Disease (EQUATOR)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The FDA declined to grant Breakthrough Therapy designation or support an Accelerated Approval pathway based on the EQUATOR study data.
Sponsor: Equillium (Industry)
Collaborators: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQ-100-02
Record Dates: First submitted 2021-10-01; First posted 2022-03-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Graft Versus Host Disease; GVHD; Acute-graft-versus-host Disease; Acute GVHD; aGVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — itolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Itolizumab (EQ001) (Experimental): Itolizumab (EQ001) administered in a blinded fashion by intravenous infusion every 2 weeks for a total of 7 doses.
  Interventions: Biological: Itolizumab
- EQ001 Placebo (Placebo Comparator): EQ001 Placebo administered in a blinded fashion by intravenous infusion every 2 weeks for a total of 7 doses
  Interventions: Drug: EQ001 Placebo

INTERVENTIONS:
Biological: Itolizumab — Itolizumab [Bmab600]
  Other Names: EQ001; Bmab600
  Arms: Itolizumab (EQ001)
Drug: EQ001 Placebo — EQ001 Placebo
  Arms: EQ001 Placebo

SUMMARY:
This is a multi-center study to compare the efficacy and safety of itolizumab versus placebo as first-line therapy for subjects with Grade III-IV aGVHD or Grade II with LGI involvement, in combination with corticosteroids

DETAILED DESCRIPTION:
This study will enroll 200 subjects at approximately 125 sites globally. Subjects will be randomized in a 1:1 ratio to active or placebo and will receive a total of 7 doses administered intravenously approximately every 2 weeks. The study follows the patients for a total of approximately 365 days.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide written informed consent/assent and to comply with all protocol procedures and assessments required for the study.
2. Is age ≥12 years and >40kg at informed consent/assent.
3. Has had an initial allogeneic HSCT for any indication using any graft source, donor source, conditioning regimen intensity or prophylaxis.
4. Has evidence of myeloid engraftment
5. Has a clinical diagnosis of aGVHD Grades III-IV or Grade II with LGI involvement based on Mount Sinai Acute GVHD International Consortium (MAGIC) grading criteria.
6. Began systemic corticosteroid treatment for aGVHD ≤72 hours prior to the start of study drug dosing AND must receive 2 mg/kg/day methylprednisolone or equivalent on Day 1.

Exclusion Criteria:

1. Evidence of morphological relapsed, progressive, persistent, or untreated malignancy, with the exception of nonmelanoma skin cancer and in situ ductal carcinoma of the breast.
2. An unplanned donor lymphocyte infusion for persistent or recurrent malignancy after HSCT.
3. Evidence of persistent molecular disease requiring treatment that was not specified prior to HSCT.
4. Evidence of cGVHD or overlap syndrome
5. Use of immunosuppressants other than corticosteroids for the treatment of aGVHD.
6. Use of any systemic corticosteroids of >0.5 mg/kg/day methylprednisolone or equivalent for any indication other than aGVHD within 7 days before the onset of aGVHD.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of itolizumab versus placebo as initial therapy for aGVHD in combination with corticosteroids in achieving early disease response. | Day 29
  Complete response at Day 29

SECONDARY OUTCOMES:
Evaluate the durability of response to itolizumab versus placebo as initial therapy for aGVHD in combination with corticosteroids. | Day 99
  Durable Complete Response rate from Day 29 through Day 99
Assess the impact of itolizumab versus placebo on other clinically relevant efficacy measures, | Day 29
  Overall Response Rates at Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Equillium, Inc.
Locations (118):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Loyola University Chicago, performing research at Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Northwell Health, Lake Success, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina (UNC), Chapel Hill, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Oncology Hematology in Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, LLC (SCRI), Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Royal Melbourne Hospital, East Melbourne
  - Austin Health, Heidelberg
  - Westmead Hospital, Westmead
- Belgium (7):
  - ULB - Institut Jules Bordet; department of Hematology, Anderlecht
  - ZNA Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Cliniques Universitaires Saint-Luc; Hematology Department, Brussels
  - UZ Leuven - Campus Gasthuisberg - Department of Hematology, Leuven
  - CHU de Liege - Hematology Department, Liège
  - AZ Delta, Roeselare
- Canada (5):
  - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center - Research Institute, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- France (13):
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - CHU de Caen - Hopital Femme-Enfant-Hematologie (FEH), Caen
  - CHU de Grenoble Hôpital Michallon, Grenoble
  - CHU de Lille - Hopital Claude Huriez, Lille
  - CHU de Nantes - Hôtel-Dieu, Lyon
  - Institut Paoli Calmettes - Hematology, Marseille
  - CHU Nice, Hospital l'Archet, Nice
  - AP-HP Hopital Saint-Louis, Paris
  - CHU Bordeaux - Hopital Haut-Leveque - Centre François Magendie, Pessac
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes Hôpital Pontchaillou, Rennes
  - CHU Toulouse, Hematology, Toulouse
  - Institut Gustave Roussy - Hematology, Villejuif
- Germany (9):
  - Charité Universitätsmedizin Berlin, Tumorimmunologie Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Koeln (AoeR), Cologne
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Martin Luther Universitat Halle-Wittenberg, Halle
  - Universitätsklinikum Jena, Jena
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitaetsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Medizinische Klinik II, Würzburg
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center Ein Karem, Jerusalem
  - Bone Marrow Transplantation Unit Rabin MC, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (11):
  - Dipartimento Malattie oncologiche ed ematologiche - U.O. Ematologia - Programma dipartimentale Terapie cellulari avanzate, Bologna, BO
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico-San Marco- Presidio Ospedaliero Ferrarotto Alessi, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli", Reggio Calabria
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - Istituto Clinico Humanitas, Rozzano
  - AOU Citta della Salute e della Scienza di Torino - Ospedale Regina Margherita, Torino
  - Azienda Ospedaliera - Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Starship Children's Hospital, Auckland, New Zealand
- Portugal (2):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, E.P.E., Porto
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Clinic Barcelona, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra - Pamplona, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marques de Valdecilla, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

REFERENCES:
- See also: Company website — https://equilliumbio.com/